CLINICAL TRIAL: NCT00049660
Title: A Randomized Phase II-III Trial Evaluating the Efficacy of Capecitabine and Vinorelbine in Anthracycline and Taxane Pre-Treated Metastatic Breast Cancer
Brief Title: Capecitabine Compared With Vinorelbine in Treating Women With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-10001-160010; EORTC-10001; EORTC-16001O; IDBBC-EORTC-10001
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Vinorelbine

INTERVENTIONS:
Drug: capecitabine
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if capecitabine is more effective than vinorelbine in treating metastatic breast cancer.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of capecitabine with that of vinorelbine in treating women who have metastatic breast cancer that has been previously treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: Phase II Study:

* Compare the response rate in women with previously treated metastatic breast cancer treated with capecitabine vs vinorelbine.
* Compare the duration of response in patients treated with these drugs.

Phase III Study:

* Compare overall and progression-free survival in patients treated with these drugs.
* Compare time to treatment failure in patients treated with these drugs.
* Compare overall safety of these drugs in these patients.
* Compare quality of life and clinical benefit response in patients treated with these drugs.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and taxane resistance (refractory vs resistant vs sensitive).

* Phase II: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive vinorelbine IV on days 1 and 8. Courses repeat every 21 days.
  * Arm II: Patients receive oral capecitabine twice daily on days 1-14. Courses repeat every 21 days.

In both arms, treatment continues in the absence of progression or unacceptable toxicity.

If sufficient response rate is determined in phase II, the phase III study is initiated.

* Phase III: Patients are randomized and receive treatment as in phase II. Quality of life is assessed prior to randomization, at weeks 3, 6, 9, 18, 24, and 30, and then every 12 weeks until disease progression.

Clinical benefit response is assessed daily while patient is on study.

Patients are followed every 6 weeks until disease progression and then every 12 weeks thereafter.

PROJECTED ACCRUAL: A total of 72 patients (36 per treatment arm) will be accrued for phase II of this study and a total of 406-452 patients (203-226 per treatment arm) will be accrued for phase III of this study within 18.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer
* Metastatic disease
* Prior treatment with taxanes in the metastatic, adjuvant, or neoadjuvant setting

  * Taxane-resistant disease allowed regardless of duration of prior therapy NOTE: Resistant disease defined as progression during or within 12 weeks after taxane therapy for metastatic disease or a disease-free interval of less than 12 months after neoadjuvant or adjuvant therapy with a taxane
  * Taxane-sensitive disease allowed if at least 4 prior courses were received NOTE: Sensitive disease defined as progression occurring more than 12 weeks after taxane therapy for metastatic disease or more than 12 months after neoadjuvant or adjuvant therapy with a taxane
* Prior treatment with anthracyclines for metastatic disease or as adjuvant treatment OR medical contraindication to treatment with anthracyclines
* At least one unidimensionally measurable lesion (phase II study)
* No CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN (5 times ULN if liver metastases present)

Renal

* Creatinine clearance greater than 50 mL/min

Cardiovascular

* No symptomatic ventricular arrhythmias
* No clinically significant congestive heart failure
* No clinical or ECG evidence of myocardial infarction within the past 12 months
* No significant coronary artery disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior malignancy within the past 5 years except contralateral breast cancer, nonmelanoma skin cancer, and adequately treated carcinoma in situ of the cervix
* No known or prior sensitivity to fluoropyrimidines, including fluorouracil
* No pre-existing grade 2 or greater neurotoxicity
* No known malabsorption or upper gastrointestinal abnormalities that would affect absorption of study drug
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy

Chemotherapy

* See Disease Characteristics
* No more than 2 prior chemotherapy lines for metastatic disease
* No prior capecitabine, vinca alkaloids, or continuous fluorouracil
* No other concurrent chemotherapy

Endocrine therapy

* Prior hormonal therapy allowed
* No concurrent hormonal therapy

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* Bisphosphonate therapy for treatment and prevention of bony metastases allowed if initiated prior to study
* No other concurrent investigational treatment
* No concurrent brivudine with capecitabine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2002-09; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martine J. Piccart-Gebhart, MD, PhD, Study Chair — Jules Bordet Institute; Chris Twelves, MD, BMedSci, FRCP, Study Chair — University of Glasgow
Locations (12):
- Belgium (4):
  - Ziekenhuis Network Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- France (2):
  - Institut Bergonie, Bordeaux
  - Centre Henri Becquerel, Rouen
- Klinikum Nuernberg - Klinikum Sued, Nurberg, Germany
- Institute of Oncology - Ljubljana, Ljubljana, Slovenia
- United Kingdom (4):
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Western Infirmary, Glasgow, Scotland

REFERENCES:
- [Result] Pajk B, Cufer T, Canney P, Ellis P, Cameron D, Blot E, Vermorken J, Coleman R, Marreaud S, Bogaerts J, Basaran G, Piccart M. Anti-tumor activity of capecitabine and vinorelbine in patients with anthracycline- and taxane-pretreated metastatic breast cancer: findings from the EORTC 10001 randomized phase II trial. Breast. 2008 Apr;17(2):180-5. doi: 10.1016/j.breast.2007.09.002. Epub 2007 Oct 31. PMID 17976988
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241